CLINICAL TRIAL: NCT01363401
Title: An Open-label, Phase I/II Trial for Safety and Efficacy Study of Autologous Bone Marrow Derived Stem Cell Treatment in Amyotrophic Lateral Sclerosis
Brief Title: Safety and Efficacy Study of Autologous Bone Marrow Derived Stem Cell Treatment in Amyotrophic Lateral Sclerosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Corestemchemon, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HYNR_CS_ALS201
Record Dates: First submitted 2011-05-30; First posted 2011-06-01 (Estimated); Results first posted 2016-07-20 (Estimated); Last update posted 2022-03-17 (Actual); Status verified 2018-09

CONDITIONS: Amyotrophic Lateral Sclerosis; ALS
Keywords: Amyotrophic lateral sclerosis; ALS; Motor neuron disease; MND; HYNR-CS inj; Autologous bone marrow derived stem cell; Intrathecal injection
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Motor Neuron Disease | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test group (Experimental): Treatment group with HYNR-CS inj.
  Interventions: Biological: HYNR-CS inj
- Control group (Experimental): No treatment with HYNR-CS inj.
  Interventions: Other: Control group

INTERVENTIONS:
Biological: HYNR-CS inj — Intrathecal injection with 1ml/10kg of body weight at an interval of 26 days.
  Arms: Test group
Other: Control group — No treatment of HYNR-CS inj
  Arms: Control group

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of autologous bone marrow-derived stem cells("HYNR-CS inj"), through intrathecal delivery for the treatment in patients with ALS.

This study consists of 2 steps. First step is a safety study of the intrathecal(IT) injection of "HYNR-CS inj" in 8 patients with ALS. In this phase 1 study, AE, laboratory test, physical examination, vital signs, Electrocardiogram, and Chest X-Ray examination were evaluated in terms of safety.

Second step is to compare the efficacy and safety between test group and control group of total 64 patients with ALS.

DETAILED DESCRIPTION:
Amyotrophic lateral sclerosis is a progressive neurodegenerative disease characterized by motor neuron loss. Despite of many trials for disease-modifying, no treatment has so far changed natural course of disease.

We have performed the pre-clinical and clinical studies using autologous bone marrow-derived stem cells in ALS. We could get the evidence that autologous bone marrow-derived stem cells have dose-dependent effects on SOD1 mice via intrathecal injection. In our results of clinical trial, intrathecal injection of autologous bone marrow-derived stem cells could slow down disease progression and might be used as a disease modifying strategy in patients with ALS.

This study was designed as a single center, randomized, open-label, parallel-group, 2-stage study, and targeted at patients diagnosed with Amyotrophic Lateral Sclerosis(Lou Gehrig's disease). The study consisted of Stage-1 study for safety evaluation and Stage-2 study for efficacy and safety evaluation of the study drug, and at Stage 1, 7 subjects eligible for the inclusion/exclusion criteria received safety evaluation for 28 days of study drug administration in twice under the protocol, and then followed Stage 2. To decide whether the study can be proceeded in 2 stages, ADR(CTCAE Version 3.0, ≥grade 3) should not appear in initial 7 subjects.

Data obtained from subjects of this study were analyzed into three: Safety Analysis, ITT(Intent-To-Treat) Analysis, and PP(Per Protocol) Analysis. However, in case of phase 1, only safety analysis was conducted, and in case of phase 2, all of safety, ITT, and PP analyses were conducted.

For ITT Analysis, all the subjects whose data on primary efficacy endpoint could be obtained following the administration of investigational drug were analyzed in analysis among subjects who were administered the investigational drug once at least. Also, Modified ITT Analysis, including 7 subjects at Stage 1, was carried out.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 25 and 75 years old
* Patients who have both signs of lower motor neuron(LMN) and upper motor neuron(UMN) degeneration by clinical, electrophysiological or neuropathologic examination
* Patients diagnosed as 'Probable' or 'Definite' ALS according to the World Federation of Neurology El Escorial criteria
* Patients who have taken Rilutek at stable background dose from 3 months ago at least before screening entry
* Patients whose duration of disease is within 5 years from the first diagnosis
* Patients with ALSFRS-R score within 31 to 46 at screening
* Patients who can visit to a hospital by walk personally or by protector's help
* Patients who provide the written consent by oneself or his/her legal representative

Exclusion Criteria:

* Patients who doesn't appropriate to the diagnostic criteria of ALS
* Patients who are diagnosed as primary lateral sclerosis(PLS) or progressive muscular atrophy(PMA)
* Patients suspected of adverse effect after stem cell injection(patients suspected of malignant tumor, risk group of psychogenic shock, patients with serious hypertension)
* Patients with ALSFRS-R score below 30 at screening
* Patients performed ventilator or tracheostomy at screening
* Patients performed gastrostomy at screening
* Patients unable to assess the efficacy of this clinical trial due to unattainable PFT(Pulmonary Functional Test) or patients with suspected 40% or less of FVC at screening
* Patients with finding of myocardial infarction or angina pectoris according to ECG, patients who have been performed Stenting or Bypass operation at screening
* Patients who have taken any other drug for clinical trial within the past 3 months at screening entry
* Patients with epilepsy
* Patients with severe renal dysfunction(serum creatinine≥2.0mg/dl)
* Patients with severe liver dysfunction(ALT, AST, bilirubin≥upper limit of normal X 2)
* Pregnant woman, lactating woman, female patients who has a pregnancy planning or who doesn't agree with adoption of contraception methods proper medically, male patients who doesn't agree with adoption of contraception methods proper to his partner during participating this study
* Patients with hemorrhagic tendency at screening
* Patients with virus infection at screening
* Patients with a known history of hypersensitivity/allergy to penicillin and streptomycin
* Patients with previous stem cell therapy
* Patients diagnosed with cancer
* Patients who have taken any drug thag can effect to bone marrow function
* Patients with any other neurological disease except ALS
* Patients with psychotic diseases

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2011-02; Primary Completion 2013-05 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Seung Hyun Kim, M.D., Ph.D., Principal Investigator — Hanyang University
Locations (1):
- Hanyang University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim H, Kim HY, Choi MR, Hwang S, Nam KH, Kim HC, Han JS, Kim KS, Yoon HS, Kim SH. Dose-dependent efficacy of ALS-human mesenchymal stem cells transplantation into cisterna magna in SOD1-G93A ALS mice. Neurosci Lett. 2010 Jan 14;468(3):190-4. doi: 10.1016/j.neulet.2009.10.074. Epub 2009 Oct 29. PMID 19879334
- [Background] Choi MR, Kim HY, Park JY, Lee TY, Baik CS, Chai YG, Jung KH, Park KS, Roh W, Kim KS, Kim SH. Selection of optimal passage of bone marrow-derived mesenchymal stem cells for stem cell therapy in patients with amyotrophic lateral sclerosis. Neurosci Lett. 2010 Mar 19;472(2):94-8. doi: 10.1016/j.neulet.2010.01.054. Epub 2010 Feb 1. PMID 20117176
- [Background] Kim HY, Kim H, Oh KW, Oh SI, Koh SH, Baik W, Noh MY, Kim KS, Kim SH. Biological markers of mesenchymal stromal cells as predictors of response to autologous stem cell transplantation in patients with amyotrophic lateral sclerosis: an investigator-initiated trial and in vivo study. Stem Cells. 2014 Oct;32(10):2724-31. doi: 10.1002/stem.1770. PMID 24966156
- [Result] Oh KW, Moon C, Kim HY, Oh SI, Park J, Lee JH, Chang IY, Kim KS, Kim SH. Phase I trial of repeated intrathecal autologous bone marrow-derived mesenchymal stromal cells in amyotrophic lateral sclerosis. Stem Cells Transl Med. 2015 Jun;4(6):590-7. doi: 10.5966/sctm.2014-0212. Epub 2015 May 1. PMID 25934946
- [Result] Oh KW, Noh MY, Kwon MS, Kim HY, Oh SI, Park J, Kim HJ, Ki CS, Kim SH. Repeated Intrathecal Mesenchymal Stem Cells for Amyotrophic Lateral Sclerosis. Ann Neurol. 2018 Sep;84(3):361-373. doi: 10.1002/ana.25302. Epub 2018 Aug 31. PMID 30048006
- See also: Corestem Inc. — http://www.corestem.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between March 2011 to May 2013, Of 10 subjects who consented to participate in the Stage 1 study, 2 subjects failed in screening, and 8 subjects were enrolled in the study. Among 71 subjects who consented to participate in the Stage 2 study, 7 subjects failed in screening, and 64 subjects were randomized.
Pre-assignment Details: Phase 1 : March 17, 2011 to November 24, 2011 Phase 2 : December 5, 2011 to May 6, 2013 The study consisted of stage 1 for safety evaluation and stage 2 for efficacy and safety evaluation of the study drug, and at stage 1, safety evaluation of the study drug, and at stage 1, safety evaluation for 28 days and then they followed stage 2.
Groups:
- HYNR-CS Inj.: Treatment group with HYNR-CS inj.
  intrathecal injection with 1ml/10kg of body weight administer twice at an interval of 26day.
- No Treatment: No treatment with HYNR-CS inj.
Period: Overall Study
Arm/Group | HYNR-CS Inj. | No Treatment
Started | 41 (Including 8 subjects of Phase 1 safety assessment. (Called "Modified ITT" in this clinical trials)) | 31
Completed | 39 | 27
Not Completed | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- No Treatment: No treatment with HYNR-CS inj.
  Take each 50mg 1 hour before a meal or 2 hours after a meal at least at an interval of 12 hours, 28 weeks(12 weeks of run-in phase plus 16 weeks of treatment phase)
- Total: Total of all reporting groups
Arm/Group | HYNR-CS Inj. | No Treatment | Total
Number analyzed (Participants) | 41 | 31 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.59 (8.59) | 52.65 (8.93) | 52.61 (8.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 18 | 35
  Male | 24 | 13 | 37
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 41 | 31 | 72
Riluzole use [Number; unit: participants]
  on Riluzole | 41 | 31 | 72
  Not on Riluzole | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: The Difference in the Changes of Amyotrophic Lateral Sclerosis Functional Rating Scale - Revised (ALSFRS-R) Between Treatment Groups and Control Groups.
Description: ALSFRS-R is ordinal rating scale questionnaire (rating 0-4 for each question, 4 is most functional, 0-48 total) of 12 functional activities. The most functional total score is 48. ALSFRS-R was evaluated at baseline and week 28.(The first injection was performed at 0 week) ALSFRS-R total score variation baseline(Visit 5) and week 16(Visit 9)
Time Frame: baseline(Visit 5) and week 16(Visit 9)
Population: The ALSFRS-R score was assessed by all the subjects in Phase 1/2 clinical trials.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HYNR-CS Inj. | No Treatment
Number analyzed (Participants) | 39 | 27
score on a scale | -1.36 (2.39) | -4.67 (3.25)

2. Secondary Outcome: Change in Appel Scale
Description: To evaluate the disease change, Appel scale will be assessed. Appel scale is a test tool, which is devised to evaluate the functional condition and variation of ALS(Lou Gehrig's disease) patients (rating 6 to between 30 and 36 points for each of 5 functional conditions, 30-164 total).
  The higher the total score presents more severe disability. This was done at Visit 1, Visit 5 and Visit 9 (week -12,0,16). The first injection was performed at 0 week(Visit 5) Appel scale total score variation baseline(Visit 5) and week 16(Visit 9)
Time Frame: baseline(Visit 5) and week 16(Visit 9)
Population: Apple scale was assessed except Two participants of No treatment group, because 1) ICU admissions for breathing therapy 2) Patients reject the measurement.
Measure: Mean (Standard Deviation); unit: point
Arm/Group | HYNR-CS Inj. | No Treatment
Number analyzed (Participants) | 39 | 25
point | 8.97 (9.24) | 17.96 (11.78)

3. Secondary Outcome: Change in Forced Vital Capacity (FVC) (Percent of Predicted Normal)
Description: Secondary efficacy was measured by comparing the rate of decline of mean FVC by treatment group.
  FVC which is a clinical scale to observe variation in patient's respiratory competence, was conducted at Visit 1, Visit 5 and Visit 9. (week -12,0,16) The first injection was performed at 0 week. FVC variation baseline(Visit 5) and week 16(Visit 9)
Time Frame: baseline(Visit 5) and week 16(Visit 9)
Population: One of the test group, FVC was assessed except because received tracheostomy during the clinical trial.
  FVC was assessed except Two participants of no treatment group because 1) ICU admissions for breathing therapy 2) Patients reject the measurement
Measure: Mean (Standard Deviation); unit: percent of prediceted
Arm/Group | HYNR-CS Inj. | No Treatment
Number analyzed (Participants) | 38 | 25
percent of prediceted | -10.51 (9.52) | -10.75 (8.40)

4. Secondary Outcome: Change in SF-36 (The Short Form (36) Health Survey is a 36 Item)
Description: The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score presents more severe disability. The higher the score presents less disability.
  This was measured at Visit 5 and Visit 9. (week 0,16) The first injection was performed at 0 week.
  The score variation baseline(Visit 5) and week 16(Visit 9)
Time Frame: baseline(Visit 5) and week 16(Visit 9)
Population: The SF-36 was assessed except Two participants of no treatment group, because 1) ICU admissions for breathing therapy 2) Patients reject the measurement.
Measure: Mean (Standard Deviation); unit: point
Arm/Group | HYNR-CS Inj. | No Treatment
Number analyzed (Participants) | 39 | 25
point | -8.59 (12.39) | -11.83 (11.28)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected for the duration of the study period: March 2011 to May 2013. Each subject was followed for AEs from consent signing to the end of their study participation.
Description: Adverse event(AE) means undesirable and unintended sign(e.g. abnormal laboratory test value) or symptom, or disease which appears following Investigational Drug use, and it shall not have causal relationship with the drug, necessarily.
  And then result of adverse events includes all the adverse events observed in 1/2 clinical trials.
Arm/Group | HYNR-CS Inj. | No Treatment
Serious Adverse Events (participants affected / at risk) | 3/41 | 3/31
Other Adverse Events (participants affected / at risk) | 28/41 | 22/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HYNR-CS Inj. (N=41) | No Treatment (N=31)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Contusion, Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HYNR-CS Inj. (N=41) | No Treatment (N=31)
Influenza like illness (General disorders) | 8 (11) | 7 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (16) | 0 (0)
Constipation (Gastrointestinal disorders) | 4 (4) | 2 (2)
Headache (Nervous system disorders) | 4 (5) | 2 (3)
Gingivitis (Infections and infestations) | 1 (1) | 0 (0)
Hepatobiliary disorders (Hepatobiliary disorders) | 3 (3) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Conjunctival disorder (Eye disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Cerumen impaction (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Wisdom teeth removal (Surgical and medical procedures) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (2) | 0 (0)
Reproductive system and breast disorders (Reproductive system and breast disorders) | 1 (2) | 0 (0)
Foreign body sensation in eyes (Eye disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 5 (6) | 1 (1)
Pain (General disorders) | 3 (4) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Coccydynia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 4 (4) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Periodontitis (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 1 (2) | 0 (0)
Tinea pedis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Vaginitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Reflux larngitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (3) | 0 (0)
Blood cholesterol increased (Investigations) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 2 (2)
Sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 (2) | 0 (0)
Hepatitis toxic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 1 (2) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (5) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No